CLINICAL TRIAL: NCT02906553
Title: The Role of Nitric Oxide in Cognition in Schizophrenia; The NOC Study (Nitric Oxide in Cognition)
Brief Title: The Role of Nitric Oxide in Cognition in Schizophrenia
Acronym: NOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16/LO/1102
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Nitric Oxide; Cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glyceryl Trinitrate (Experimental): Glyceryl Trinitrate, sublingual spray, 3 x 0.4mg dose, once per day for 3 days in total.
  Interventions: Drug: Glyceryl Trinitrate
- Placebo (Placebo Comparator): The formulation composition of the placebo will be the same as the active spray minus the Glyceryl Trinitrate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glyceryl Trinitrate
  Arms: Glyceryl Trinitrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the role of the Nitric Oxide system in cognition in patients with schizophrenia. Participants will be randomised to 2 equal groups and receive either the Nitric Oxide donor molecule glyceryl trinitrate, or a placebo. Performance on several cognitive tasks will be assessed.

DETAILED DESCRIPTION:
Nitric oxide [NO] is a gaseous neurotransmitter substance found in the brain. Nitric oxide is integrated with the glutamate system. Glutamate has received considerable attention as an important factor in the cognitive distortions and cognitive impairments that underlie schizophrenia. Deficits in glutamate in schizophrenia may impact upon cognition via the NO system, as glutamate receptors signal by way of NO.

Here the investigators aim to extend knowledge of glutamate-NO systems by directly examining the role of NO in cognition in patients with psychosis. We aim to assess the role of the NO system in cognition, downstream of glutamate and before patients are started on any anti-psychotic medication which perturb brain neurochemistry.

The primary outcome measure is change in a particular style of cognition referred to as 'jumping to conclusions' following the administration of a potent Nitric Oxide donor molecule [glyceryl trinitrate (GTN)], under placebo-controlled, double-blind conditions. This will shed light on the direct role of NO in cognition in psychosis, beyond the glutamate system.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Patients undergoing an acute psychotic episode (defined as score > 4 on question P1 of the PANSS positive subscale) requiring full-time hospitalisation according to clinical referral by the relevant mental health service
* Demonstrates capacity and willing to give informed consent
* Female participants willing to have a pregnancy test before treatment
* Currently unmedicated with antipsychotic medication

Exclusion Criteria:

* Major physical illness
* Prior history of intolerance to glyceryl trinitrate
* Homicidal or suicidal
* Pregnant or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The emotionally salient version of the Jumping to Conclusions (JTC) task | Change in performance from baseline to Day1, Day 2, Day 3, Day 7

SECONDARY OUTCOMES:
The Hopkins Verbal Learning Task - Revised, immediate recall | Change from baseline to Day1, Day 2, Day 3, Day 7
Positive and negative syndrome scale (PANSS) (videotaped) | Change from baseline to Day1, Day 2, Day 3, Day 7
The Bond-Lader Visual Analog Scales | Change from baseline to Day1, Day 2, Day 3, Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Paul Morrison, MRCPsych, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merritt K, Catalan A, Cowley S, Demjaha A, Taylor M, McGuire P, Cooper R, Morrison P. Glyceryl trinitrate in first-episode psychosis unmedicated with antipsychotics: A randomised controlled pilot study. J Psychopharmacol. 2020 Aug;34(8):839-847. doi: 10.1177/0269881120922967. Epub 2020 May 21. PMID 32436761